CLINICAL TRIAL: NCT05097716
Title: PHASE 1, OPEN-LABEL, FIXED-SEQUENCE, 2-PERIOD STUDY TO ESTIMATE THE EFFECT OF MULTIPLE-DOSE RITLECITINIB (PF-06651600) ON THE PHARMACOKINETICS OF SINGLE-DOSE TOLBUTAMIDE IN HEALTHY PARTICIPANTS
Brief Title: Study to Evaluate the Effect of Multiple-Dose Ritlecitinib on the Pharmacokinetics (PK) of Tolbutamide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: B7981069
Record Dates: First submitted 2021-10-14; First posted 2021-10-28 (Actual); Results first posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2022-12

CONDITIONS: Healthy Volunteers
Keywords: pharmacokinetics (PK)
MeSH Terms: interventions — PF-06651600; Tolbutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ritlecitinib and tolbutamide (Experimental): In Period 1, participants will be dosed with a single administration of tolbutamide 500 mg tablet on Day 1. Period 1 will be immediately followed by Period 2 with no washout. In Period 2, participants will be dosed with oral 200 mg ritlecitinib QD for 10 days followed by administration of a single dose of 500 mg tolbutamide oral tablet within approximately 5 minutes after administration of a 200 mg dose of ritlecitinib on the morning of Day 10.
  Interventions: Drug: Ritlecitinib; Drug: Tolbutamide

INTERVENTIONS:
Drug: Ritlecitinib — Ritlecitinib 200 mg provided as four 50 mg oral capsules
  Other Names: PF-06651600
Drug: Tolbutamide — Tolbutamide 500 mg provided as one 500 mg oral tablet

SUMMARY:
This is a Phase 1, 2-period, multiple-dose, open-label, single fixed sequence study of the effect of ritlecitinib on tolbutamide pharmacokinetics in healthy participants.

DETAILED DESCRIPTION:
A total of approximately 12 healthy male and/or female participants will be enrolled in the study to obtain at least 10 evaluable participants who complete the study. This is an open-label study not requiring an assessment of efficacy or pharmacodynamics markers, but it will include pharmacokinetic estimation drug-drug interactions.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female participants who are healthy as determined by medical evaluation including medical history, full physical examination (including BP and pulse rate measurements), clinical laboratory tests, and 12-lead ECG.
* BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

* Past/present clinically significant hematological, renal, endocrine, pulmonary, GI, CV, hepatic, psychiatric, neurological, dermatological or allergic disease (including drug allergies).
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* Infection with hepatitis B or C viruses.
* Participants with any of the following acute or chronic infections or infection history: any infection requiring treatment within 2 weeks prior to the start of study participation; any infection requiring hospitalization or parenteral antimicrobial therapy within 60 days of the first dose of investigational product; any infection judged to be an opportunistic infection or clinically significant within the past 6 months of the first dose of investigational product; known active or history of recurrent bacterial, viral, fungal, mycobacterial or other infections; history of recurrent localized dermatomal herpes zoster, or history of disseminated (single episode) herpes simplex or disseminated herpes zoster.
* History of any lymphoproliferative disorder such as EBV related lymphoproliferative disorder, history of lymphoma, history of leukemia, or signs or symptoms suggestive of current lymphatic or lymphoid disease.
* Known presence or a history of malignancy other than a successfully treated or excised non-metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981069

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 12 participants were enrolled in the study. All participants were treated in Period 1 (tolbutamide treatment alone). Ten participants were treated in Period 2 (multiple dose ritlecitinib plus single dose tolbutamide treatment).
Groups:
- Period 1: Tolbutamide and Period 2: Ritlecitinib + Tolbutamide: Participants in Period 1 were dosed with a single administration of tolbutamide 500 mg tablet on Day 1. Period 1 was immediately followed by Period 2 with no washout. Participants in Period 2 were dosed with oral 200 mg ritlecitinib once daily (QD) for 10 days followed by administration of a single dose of 500 mg tolbutamide oral tablet within approximately 5 minutes after administration of ritlecitinib on the morning of Day 10.
Period: Period 1
Arm/Group | Period 1: Tolbutamide and Period 2: Ritlecitinib + Tolbutamide
Started | 12
Completed | 10
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Close contact with highly-transmissible infection | 1
Period: Period 2
Arm/Group | Period 1: Tolbutamide and Period 2: Ritlecitinib + Tolbutamide
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants assigned to the study intervention.
Groups:
- Male: Male participants were healthy adults between 18-65 years of age. No contraception methods were required for male participants in this study.
- Female: Female participants were healthy adults between 18-65 years of age. A female participant was eligible to participate if she was not pregnant or breastfeeding, and at least 1 of the following conditions applied: was not a woman of childbearing potential, OR was a woman of childbearing potential using a contraceptive method that was highly effective.
- Total: Total of all reporting groups
Arm/Group | Male | Female | Total
Number analyzed (Participants) | 9 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean | 37.4 (12.57) | 48.7 (11.15) | 40.3 (12.78)
Age, Continuous [Median (Full Range); unit: Years]
  Median | 36.0 [23.0 to 57.0] | 53.0 [36.0 to 57.0] | 37.0 [23.0 to 57.0]
Age, Customized [Count of Participants; unit: Participants]
  <18 | 0 | 0 | 0
  18-44 | 6 | 1 | 7
  45-64 | 3 | 2 | 5
  >=65 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 9 | 0 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 8 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 2 | 7
  Black or African American | 4 | 0 | 4
  Asian | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Tolbutamide Administered With and Without Ritlecitinib
Description: Cmax was defined as maximum observed plasma concentration. The determination method of Cmax was observing directly from data.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, and 36 hours post-dose of tolbutamide in Period 1 (Days 1 and 2) and Period 2 (Days 10 and 11)
Population: Analysis population included all participants treated who had at least 1 concentration in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL (nanogram/milliliter)
Groups:
- Period 1: Tolbutamide: Participants in Period 1 were dosed with a single administration of tolbutamide 500 mg tablet on Day 1.
- Period 2: Ritlecitinib + Tolbutamide: Participants in Period 2 were dosed with oral 200 mg ritlecitinib QD for 10 days followed by administration of a single dose of 500 mg tolbutamide oral tablet within approximately 5 minutes after administration of ritlecitinib on the morning of Day 10.
Arm/Group | Period 1: Tolbutamide | Period 2: Ritlecitinib + Tolbutamide
Number analyzed (Participants) | 12 | 10
ng/mL (nanogram/milliliter) | 44240 (15) | 45740 (17)
Statistical Analysis 1: Comparison: Period 1: Tolbutamide vs Period 2: Ritlecitinib + Tolbutamide; Test type: Equivalence — 90% CI; ratio of adjusted geometric means = 103.01, 90% CI 2-sided [96.66 to 109.77] — The comparison was Test vs. Reference (Ritlecitinib + Tolbutamide vs. Tolbutamide)

2. Primary Outcome: Area Under the Plasma Concentration Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of Tolbutamide Administered With and Without Ritlecitinib
Description: AUCinf was defined as area under the plasma concentration time profile from time 0 extrapolated to infinite time.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, and 36 hours post-dose in Period 1 (Days 1 and 2) and Period 2 (Days 10 and 11)
Population: Analysis population included all participants treated who had at least 1 concentration in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Period 1: Tolbutamide | Period 2: Ritlecitinib + Tolbutamide
Number analyzed (Participants) | 12 | 10
ng*hr/mL | 608600 (20) | 586500 (30)
Statistical Analysis 1: Comparison: Period 1: Tolbutamide vs Period 2: Ritlecitinib + Tolbutamide; Test type: Equivalence — 90% CI; ratio of adjusted geometric means = 99.05, 90% CI 2-sided [92.01 to 106.62] — The comparison was Test vs. Reference (Ritlecitinib + Tolbutamide vs. Tolbutamide)

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) - All Causalities and Treatment Related
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation where participants were administered a product; the event needed not necessarily have a causal relationship with the treatment or usage. TEAEs were events between first dose of study drug and up to discharge from study that were absent before treatment or that worsened relative to pretreatment state. A treatment-related AE was any untoward medical occurrence attributed to the study drug in a participant who received study drug.
Time Frame: From screening up to a follow-up phone call between 28 and 35 calendar days after the last administration of the investigational product and early termination (if applicable)
Population: Analysis population included all participants assigned to the study intervention and who took at least 1 dose of the study intervention. Participants were analyzed according to the intervention they actually received.
Measure: Number; unit: Participants
Groups:
- Period 2: Ritlecitinib: Participants in Period 2 were dosed with oral 200 mg ritlecitinib QD for 10 days.
Arm/Group | Period 1: Tolbutamide | Period 2: Ritlecitinib | Period 2: Ritlecitinib + Tolbutamide
Number analyzed (Participants) | 12 | 10 | 10
Participants
  All-Causality | 1 | 2 | 2
  Treatment-Related | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From screening up to a follow-up phone call between 28 and 35 calendar days after the last administration of the investigational product and early termination (if applicable)
Description: The same event may appear as both an AE and a serious adverse event (SAE). An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Period 1: Tolbutamide | Period 2: Ritlecitinib | Period 2: Ritlecitinib + Tolbutamide
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/12 | 2/10 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: Tolbutamide (N=12) | Period 2: Ritlecitinib (N=10) | Period 2: Ritlecitinib + Tolbutamide (N=10)
Pain (General disorders) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/16/NCT05097716/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT05097716/SAP_001.pdf